CLINICAL TRIAL: NCT06082375
Title: Effect of 8-week Supplementation With Vitamin D3 on Functional and Cognitive Performance in Patients With Chronic Low Back Pain Eligible for Neurosurgery Intervention
Brief Title: Supplementation With Vitamin D3 on Chronic Low Back Pain Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Patryk Chromiec, Senior assistant professor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SVITD
Record Dates: First submitted 2023-09-27; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain; vitamin D; neurosurgery; functional; cognitive
MeSH Terms: interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental): Individually adapted to each participant based on BMI, dose of vitamin D3 in drops.
  1. BMI 19-25 - 4000 IU
  2. BMI 25-29,9- 6000 IU
  3. BMI >30- 8000 IU
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): The placebo group will receive drops containing vegetable oil in the same bottles as vitamin D3.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D3 in the form of cholecalciferol.
  Other Names: cholecalciferol
  Arms: Vitamin D
Dietary Supplement: Placebo — Vegetable oil.
  Arms: Placebo

SUMMARY:
The study was designed as a randomized double-blind placebo-controlled clinical trial with 8-week Vitamin D3 and physical activity intervention. The protocol was approved by Independent Bioethics Committee for Scientific Research at Medical University of Gdańsk (No. 525/2018), in accordance with the Declaration of Helsinki. We enrol 40 patient (aged ≥ 35), Patients diagnosed with chronic pain in the lumbar spine, qualified for surgical treatment at the Department of Neurosurgery Medicinal Unit in Gdańsk. Participation in the study was voluntary, and the condition for participation was obtaining informed consent from the patient.

DETAILED DESCRIPTION:
Before starting supplementation, a blood sample was taken from patients to determine the status of vitamin D3, measurements of hydroxylated vitamin D at position 25 (25OHD3) and monitoring of inflammatory markers such as Interleukin-6; TumorNecrosisFactor-α. This measurement was performed in the University laboratory in Gdańsk according to a standard, generally accepted method for the determination of a given compound. The blood sample was taken by a qualified nurse. This measurement was repeated to control vitamin D levels and markers of inflammation:

* After 6 weeks of supplementation (before surgery);
* After 2 weeks of supplementation (after surgery);

Patients was supplemented with vitamin D or placebo for 6 weeks before surgery and was continue supplementation for 6 weeks after surgery. According to the value of the Body Mass Index, the dose of vitamin D will be appropriately selected for each group:

* Group 1 BMI 19-25 - 4000 IU
* Group 2 BMI 25-29,9- 6000 IU
* Group 3 BMI >30- 8000 IU

A person was appointed to coordinate the allocation of patients to the two groups. Patients was not informed whether they are receiving vitamin D or a placebo. The treating doctors, radiology specialists and the rest of the team was not know what group the patient is in. Within individual groups, patients was randomly assigned to:

* Group A - patients supplemented with placebo;
* Group B - patients supplemented with vitamin D3; Patients was informed about the purpose of the research and was receive. The patients diet was monitored during supplementation by a certified clinical dietitian using food diaries. The food diary is a basic tool for monitoring the diet of test subjects. After appropriate training, the respondents are able to fill in the diary on their own, writing down all the meals eaten during the day and snacks with drinks. It is a qualitative and quantitative method that allows you to analyze the diet so far and draw appropriate conclusions.

Patients from both groups who will not have contraindications to exercise, 2 weeks after surgery, was divided into a group for 6 weeks of home routine physical activity and a group not doing any additional physical activity.

* Group A1 - placebo supplementation + exercise
* Group A2 - placebo supplementation + no exercise
* Group B1 - supplementation with vit. D + exercises
* Group B2 - supplementation with vit. D + no exercise

ELIGIBILITY:
Inclusion Criteria:

* Pain in the lumbar spine that lasts more than 6 months (diagnosed by signs and symptoms, and tests such as magnetic resonance imaging (MRI));
* Failure to respond to medications and physical therapies;
* Visual Analog Pain Scale (VAS), (0-100) score greater than or equal to 50;
* Numerical Rating Scale (NRS);

Exclusion Criteria:

* Rheumatoid arthritis;
* Diagnosed mental illness;
* Drugs;
* Metabolic bone diseases (hypo or hyperparasitism);
* Chronic kidney diseases and diseases affecting vitamin D metabolism (stomach surgery, chronic liver diseases, kidney failure, malabsorption disorders, systemic infection, tumors, etc.)
* Medicines that alter the metabolism of bones such as corticosteroids or bisphosphonates;
* Vitamin D supplements in the last 3 months;
* BMI: less than 19;

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in vitamin D3 status at blood serum | Baseline and Week 8
  Blood sample will be taken from patients to determine the status of vitamin D3, measurements of hydroxylated vitamin D at position 25 (25OHD3)
Change in vitamin Interleukin-6 status at blood serum | Baseline and Week 8
  Blood sample will be taken from patients to determine the status of interleukin-6, measurements to show changes in inflammation in the blood.
Change in vitamin TumorNecrosisFactor-alfa status at blood serum | Baseline and Week 8
  Blood sample will be taken from patients to determine the status of Tumor Necrosis Factor, measurements to show changes in inflammation in the blood.
Change in cognitive test Quality of life Short Form-36 questionnaire | Baseline and Week 8
  Validated cognitive tests assessing patients' quality of life. The Short Form - 36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health or emotional wellbeing
Change in cognitive test Chalder Fatigue Questionnaire | Baseline and Week 8
  Validated cognitive tests assessing patients' quality of life.
  The subject answers the questions using a 4-step scale (choosing between "better than usual," "no more than usual," "worse than usual" and "much worse than usual"). Answers to the first 7 items give an insight into the intensity of the physical fatigue and the next 4 give a picture of the mental fatigue. The overall score is obtained by adding all the items. There are 2 scoring systems:
  * a Likert system, where the subject's answers are evaluated by awarding 0, 1, 2 or 3 pts, giving a maximum of 33 pts;
  * a bimodal system, which ignores the severity of responses and categorizes the answers as a "problem" ("more than usual" and "much more than usual" - 1 pt) or "no problem" ("less than usual" and "no more than usual" - 0 pt), giving a maximum of 11 pts.
Change in functional test Up&Go | Baseline and Week 8
  Up&Go Test aimed at checking the task completion time as a functional element. Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
  For password: "Go," the patient begins:
  1. Stand up from the chair. 2. Walk to the line on the floor at your normal pace.
  3. Turn. 4. Walk back to the chair at your normal pace. 5. Sit down again. On the word "Go," begin timing. Stop timing after patient sits back down. Record time: time in Seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kaczor, Professor, Study Chair — Medical University of Gdansk
Locations (1):
- Medical University, Gdansk, Pomeranian Voivodeship, Poland